CLINICAL TRIAL: NCT02140138
Title: An Open Label Randomised Phase II Trial of RNActive® Cancer Vaccine (CV9104) in High Risk and Intermediate Risk Patients With Prostate Cancer
Brief Title: An Open Label Randomised Trial of RNActive® Cancer Vaccine in High Risk and Intermediate Risk Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was terminated after enrolment of 35 instead of 36 evaluable patients for administrative reasons.
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV-9104-007; 2013-004489-32 (EudraCT Number)
Record Dates: First submitted 2014-04-07; First posted 2014-05-16 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (i.d. vaccinations with needle free injection device) (Experimental): Duration: Patients in Arm A will receive a total of 4 vaccinations with CV9104 in weeks 1, 2, 3 and 5. These patients will undergo radical prostatectomy at least 1 week but not later than 2 weeks after the 4th vaccination (week 6 or 7). After surgery high risk or very high risk patients will be offered to receive 2 additional vaccinations with CV9104 at week 8 and 10 post surgery.
  Administration: At each vaccination visit each of the 6 components of CV9104 vaccine will be injected individually, divided in two separate intradermal injections. These 12 Injections will be distributed over the 4 limbs (3 injections in each upper arm and thigh).
  Administration site: Skin of the lateral parts of the upper arms (over the deltoid regions) and the lateral part of the thighs.
  Dose: 2 x 80 μg mRNA per injection (2 x 100 μL), equals 160 μg mRNA per RNActive® drug product component
  Interventions: Biological: CV9104; Device: needle free injection device (Tropis®)
- Arm B (i.d. vaccination by conventional injection) (Experimental): Duration: Patients in Arm B will receive a total of 4 vaccinations with CV9104 in weeks 1, 2, 3 and 5. These patients will undergo radical prostatectomy at least 1 week but not later than 2 weeks after the 4th vaccination (week 6 or 7). After surgery high risk or very high risk patients will be offered to receive 2 additional vaccinations with CV9104 at week 8 and 10 post surgery.
  Administration: At each vaccination visit each of the 6 components of CV9104 vaccine will be injected individually, divided in two separate intradermal injections. These 12 Injections will be distributed over the 4 limbs (3 injections in each upper arm and thigh).
  Administration site: Skin of the medial part of the upper arms and thigh
  Dose: 2 x 160 μg mRNA per injection (2 x 200 μL), equals 320 μg mRNA per RNActive® drug product component
  Interventions: Biological: CV9104
- Arm C (i.d. vaccination with needle free injection device) (Other): Duration: Patients in Arm C will receive no vaccination before radical prostatectomy. After surgery high risk or very high risk patients will be offered to receive 6 vaccinations with CV9104 at week 8, 9, 10, 12, 14 and 16 after surgery.
  Administration: At each vaccination visit each of the 6 components of CV9104 vaccine will be injected individually, divided in two separate intradermal injections. These 12 Injections will be distributed over the 4 limbs (3 injections in each upper arm and thigh).
  Administration site: Skin of the lateral parts of the upper arms (over the deltoid regions) and the lateral part of the thighs.
  Dose: 2 x 80 μg mRNA per injection (2 x 100 μL), equals 160 μg mRNA per RNActive® drug product component
  Interventions: Biological: CV9104; Device: needle free injection device (Tropis®)

INTERVENTIONS:
Biological: CV9104
Device: needle free injection device (Tropis®)
  Arms: Arm A (i.d. vaccinations with needle free injection device); Arm C (i.d. vaccination with needle free injection device)

SUMMARY:
The purpose of this study is to evaluate the induction of immune responses against CV9104 administered by conventional intradermal injection or with a needle-free intradermal injection device and to assess the safety and tolerability of CV9104 administered by conventional intradermal injection versus injection with a needle-free intradermal injection device versus no injection.

DETAILED DESCRIPTION:
This study is the second clinical trial of the RNActive® vaccine. It is composed of 6 RNActive® drug product components, coding for 6 antigens that are overexpressed in PCA compared to healthy tissue. Each of the 6 prostate specific antigens that are encoded by CV9104 are capable of inducing adaptive immunity.

Needle-free injection systems, like the Tropis® device for i.d. injection, overcome the disadvantages related to needle- and syringe-based i.d. injections. Tropis® is currently used in different vaccine clinical trials around the world. The use of Tropis® for i.d. delivery of CV9104 has been approved by BfArM.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged ≥18 years
2. Histologically confirmed adenocarcinoma of the prostate with at least one of the following criteria for intermediate to high risk disease:

   * Gleason Score 7-10
   * Serum PSA > 10 ng/mL
   * cT2b-c / cT3a without tumor fixation to adjacent organs
3. Absence of very high risk or metastatic disease (i.e. cT3b-T4 N0 or any T, N1 or M1) confirmed by EITHER CT or MRI of the abdomen and pelvis (in patients with a Gleason score ≥ 8 or a clinical stage T3) and bone scintigraphy (in patients with a PSA of ≥ 10 ng/mL, a Gleason score ≥ 8, a clinical stage T3 or bone pain or other symptoms of metastatic disease)
4. Patient is physically fit and eligible for radical prostatectomy based on best clinical evidence and has already decided to undergo radical prostatectomy after discussion of potential alternative treatment options.
5. ECOG 0 or 1
6. No prior treatment for prostate cancer including prior surgery (including TURP), pelvic lymph node dissection, radiation therapy, antihormonal therapy or chemotherapy
7. Adequate organ function:

   * Bone marrow function: hemoglobin ≥ 12 g/dL; white blood cell count (WBC) ≥ 3.0 x 109/L; lymphocyte count ≥ 1.0 x 109/L; absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count ≥ 150 x 109/L
   * Hepatic: AST, ALT and GGT ≤ 2.5 times upper limit of normal (ULN); bilirubin ≤ 1.5 x ULN
   * Renal: creatinine ≤ 2 mg/dL and creatinine clearance ≥ 45 mL/min/1.73 m2
8. Fertile men and their female partners must use a highly effective method of contraception resulting in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Those methods include implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs) or abstinence. The contraception should be applied from enrollment until 4 weeks after the last vaccination.
9. Written informed consent must be obtained prior to conducting any study-specific procedures.

Exclusion Criteria:

1. Concurrent treatment with systemic steroids or other immunosuppressive agents [except topical (inhaled, topical, nasal) and replacement therapy for adrenal insufficiency] should be strictly avoided throughout the study, concomitant treatment with immunomodulating agents including herbal remedies (e.g. mistletoe extract) has to be avoided during study treatment and must be discontinued at least 28 days prior to the start of treatment
2. Previous therapies with investigational anticancer agents including cancer vaccines or other cancer immunotherapies
3. Prior splenectomy
4. Prior allogeneic bone marrow transplant
5. History of autoimmune disorders such as sarcoidosis, lupus erythematosus, rheumatoid arthritis, glomerulonephritis or systemic vasculitis (except autoimmune thyroiditis with only thyroid hormone replacement and stable disease > 1 year)
6. Primary or secondary immune deficiency
7. Seropositive for HIV, HBV (except after Hep B vaccination) or HCV infection
8. History of other malignancies over the last 5 years (except adequately treated basal cell or squamous cell carcinoma of the skin)
9. Uncontrolled medical condition considered as high risk for the treatment with an investigational drug including unstable diabetes mellitus, symptomatic congestive heart failure (NYHA 3 and 4); coronary heart disease with unstable angina pectoris, history of myocardial infarction, or coronary artery intervention (PTCA, stenting) within 6 months prior to enrolment; significant cardiac arrhythmia, history of stroke or transient ischemic attack. Severe hypertension according to WHO criteria or systolic blood pressure ≥ 180 mmHg at the time of enrolment.
10. History of seizures, encephalitis or multiple sclerosis
11. History of inflammatory bowel disease or Crohn´s disease or ulcerative colitis
12. Active drug abuse or chronic alcoholism
13. Active skin disease (atopic eczema, psoriasis) in the areas for vaccine injection preventing the i.d. administration of study product into areas of healthy skin
14. Allergies to any component of the study drug including known allergy to protamine sulphate (e.g. allergy to protamine containing insulins) or fish allergy.
15. Prior vasectomy
16. Known type I allergy to β-lactam antibiotics
17. Active infections (including acute prostatitis) requiring anti-infectious therapy at the time of enrolment: leucocytosis ≥ 9000/μL; CRP elevation ≥ 2.5 times upper limit of normal or leucocyturia of ≥ 75 cells/μl (equals ≥ grade 2+ on two consecutive Combur® urinalysis specimen)
18. Uncontrolled urinary retention or hydronephrosis
19. Inability to provide informed consent due to mental impairment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Induction of antigen-specific cellular and humoral immune response to the vaccine antigens. | Up to one week before the date of surgery.

SECONDARY OUTCOMES:
Incidence and severity of adverse device effects, adverse events and laboratory abnormalities, graded according to NCI-CTCAE version 4.0 criteria | From ICF signature till end of study (max. up to week 20 after first study treatment in arm A and B and up to week 26 after first study treatment in arm C)
Occurrence of serious adverse events | From ICF signature till end of study (max. up to week 20 after first study treatment in arm A and B and up to week 26 after first study treatment in arm C)
Occurrence of treatment discontinuation due to adverse events | From time of first to last study treatment
Change in PSA serum levels during the presurgical period and, in patients receiving postsurgical vaccinations, change in PSA during the postsurgical period | At screening, at baseline (week 1), at the last presurgical visit (week 6 in arm A and B, week 3-6 in arm C), at the first postsurgical visit (8 weeks after surgery) and at the end of study (max. up to week 21 in arm A and B and up to week 27 in arm C)

OTHER OUTCOMES:
Assessment of immune cell infiltration, and gene expression profiles in prostatectomy tissue samples. | tissue collection at prostatectomy (week 6-7 in arm A and B, week 4-7 in arm C)
Assessment of immune parameters and biomarkers in blood and exprimate urine | At baseline (week 1), at the last presurgical visit (week 6 in arm A and B, week 3-6 in arm C), at the first post surgical visit (8 weeks after surgery; blood only) and in week 13 after surgery (in arm C, receiving vaccinations after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Stenzl, Prof. Dr. med., Principal Investigator — Klinik für Urologie, Universitätsklinikum Tübingen
Locations (3):
- Germany (3):
  - Nationales Zentrum für Tumorerkrankungen, Medizinische Onkologie, Heidelberg, Baden-Wurttemberg
  - Klinik für Urologie, Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum rechts der Isar, Urologische Klinik und Poliklinik der Technischen Universität München, München, Bavaria